CLINICAL TRIAL: NCT04300426
Title: Aiming to Reduce Disease-related Gastrointestinal Symptoms in Systemic Sclerosis by Repeat Intestinal Infusions of Anaerobic Cultivated Human Intestinal Microbiome (ACHIM); a Randomized, Double-blind Placebo-controlled 20 Week Study
Brief Title: Safety and Efficacy of Anaerobic Cultivated Human Intestinal Microbiome Transplantation in Systemic Sclerosis (ReSScue)
Acronym: ReSScue
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Oslo University Hospital (Other)
Collaborators: South-Eastern Norway Regional Health Authority (Other); Haukeland University Hospital (Other); St. Olavs Hospital (Other); University Hospital of North Norway (Other)
Responsible Party: Principal Investigator, Anna-Maria Hoffmann-Vold, National PI, Oslo University Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2019-004400-35
Record Dates: First submitted 2020-02-25; First posted 2020-03-09 (Actual); Last update posted 2022-10-12 (Actual); Status verified 2022-10

CONDITIONS: Systemic Sclerosis
MeSH Terms: conditions — Scleroderma, Systemic | interventions — Fecal Microbiota Transplantation

STUDY DESIGN:
Intervention Model Description: The 20-week study period consists of a 12-week induction phase (Part A1), with randomized, double-blind parallel group interventions by endoscopic infusions at weeks 0 and 2, and an 8-week maintenance phase (Part A2) where all participants receive one single open label endoscopic infusion on week 12. Additionally, all participants who complete the 20-week study period are followed for a maximum 16 weeks monitoring period (Part B) to obtain longer-term data on safety and durability of intervention effects.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Masking will apply for the whole duration of study until end of study defined as week 20 visit for the last participant.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ACHIM by gastroduodenoscopy (Experimental): Intestinal microbiota (acronym ACHIM - anaerobically cultured human intestinal microbiota) will be administered by gastroduodenoscope twice (given at baseline and study-week 2). Each with volume 30 ml, containing approximately 10^9 bacteria / ml.
  Primary outcome measured at week 12. At week 12 an open label administration of ACHIM to all participants. Thereafter an 8 (+16) week period observation. Blind from the first intervention will be maintained through-out the duration of the study.
  Interventions: Drug: "ACHIM" as solute (10^9 intestinal microbes/ml)
- Placebo by gastroduodenoscopy (Placebo Comparator): ACHIM culture media (no bacteria) will be administered by gastroduodenoscope twice (given at baseline and study-week 2). Each with volume 30 ml.
  Primary outcome measured at week 12. At week 12 an open label administration of ACHIM to all participants. Thereafter an 8 (+16) week period observation. Blind from the first intervention will be maintained through-out the duration of the study.
  Interventions: Drug: "ACHIM" as solute (10^9 intestinal microbes/ml)

INTERVENTIONS:
Drug: "ACHIM" as solute (10^9 intestinal microbes/ml) — Culture of intesinal microbiota originally derived from a healthy subject are administered to a person with presumed dysbiotic intestinal symptoms with an objective to treat these symptoms.
  Other Names: Fecal microbiota transplantation

SUMMARY:
This study evaluates the effect of intestinal microbiota therapy on gastro-intestinal symptoms in patients with systemic sclerosis (SSc). This is a mulicenter randomized controlled trial conducted at university hospitals in Oslo, Tromsø, Bergen and Trondheim in Norway. In part A1, half of the patients will receive active substance (intestinal microbiota cultured in the lab - "ACHIM") in the small intestine twice by gastroduodenoscopy, the other half will receive placebo. The primary outcome will be measured on week 12 by patient reported outcome measures. In part A2, all participants receive ACHIM at week 12, with an 8 week follow-up for all. A step-wise follow-up will be done in part B up to 16 weeks after week 20 until the last participant finish week 20 visit, which is defined as end of study.The blind from the first intervention will not be opened before end of study.

ELIGIBILITY:
Inclusion Criteria:

1. Participant must be 18 to 85 years of age inclusive, at the time of signing the informed consent.
2. Participants must have been clinically diagnosed with SSc by a rheumatologist having experience with the disease.
3. Participants must have disease characteristics that fulfill the 2013 ACR/EULAR classification criteria for SSc.
4. Participants must be able to understand and follow trial procedures including completion of questionnaires regarding Patient Reported Outcome measures, such as the Norwegian version of the UCLA GIT V2.0 score.
5. Participants must have moderate to severe SSc-related lower GI symptoms at time of inclusion, as defined by UCLA GIT score values of ≥1.01 for bloating and/or ≥0.50 for diarrhea at the screening visit.
6. Male and female
7. Capable of giving signed informed consent as described in Appendix 1 which includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and in this protocol.

Exclusion Criteria:

* Medical Conditions

  1. Cardiovascular diseases, any of the following

     1. Severe hypertension, uncontrolled under treatment (≥160/100 mmHg), within 6 month of Visit 1
     2. Myocardial infarction within 6 months of Visit 1
     3. Unstable cardiac angina within 6 months of Visit 1
  2. Lung disease with impaired respiratory function, any of the following

     1. Forced Vital Capacity (FVC) < 50% of expected reference value within 12 month of Visit 1
     2. Diffusing lung capacity for carbon monoxide (DLCO) < 40% of expected reference value within 12 month of Visit 1
     3. LTOT or lung-tx
  3. Significant pulmonary hypertension, any of the following

     1. Previous clinical or echocardiographic evidence of significant right heart failure
     2. History of right heart catheterisation showing a cardiac index ≤ 2 l/min/m²
  4. History of thrombotic event (including stroke and transient ischemic attack) within 12 months of Visit 1
  5. Severe anemia with Hb < 8.0 g/l within 4 weeks prior to Visit 1. Repeat testing of Hb is allowed.
  6. Bleeding risk, any of the following

     1. History of hemorrhagic central nervous system (CNS) event within 12 months of Visit 1.
     2. Known genetic predisposition to bleeding
     3. Platelet counts < 50 x 109/l
  7. Chronic liver disease or gastro-intestinal condition, any of the following

     1. Primary biliary cholangitis
     2. Primary sclerosing cholangitis
     3. Decompensated chronic liver disease
     4. Inflammatory bowel disease
     5. Celiac disease treated for less than 12 months.
  8. Gastro-intestinal surgery performed within the within 12 months of Visit 1
  9. Hepatic dysfunction, as defined as AST, ALT or bilirubin levels >3 times the Upper limit of normal range (x ULN) within 4 weeks prior to Visit 1. Repeat testing of AST, ALT and bilirubin are allowed in participants with no prior history of hepatic dysfunction.
  10. Chronic renal insufficiency, with estimated Glomerular Filtration Rate (eGFR) < 30.
  11. Active digital ulcers within 4 weeks of Visit 1.
  12. Anaphylactic food allergy.
  13. Eating disorder diagnosed by a physician
  14. Other diseases or conditions that may interfere with testing procedures (for example inability to conduct gastroduodenoscopy) or in the judgment of the Investigator may interfere with trial participation or may put the patient at risk when participating in this trial (for example severe GI symptoms due to other diseases than SSc).

      Prior/Concomitant Therapy
  15. Any antibiotic therapy within 3 months of Visit 1
  16. Prednisone >10 mg/day or equivalent within 4 weeks prior to Visit 1
  17. Cyclophosphamide or rituximab treatment within 6 months prior to Visit 1
  18. Unstable background monotherapy with any of the following therapeutics; mycophenolate mofetil/sodium, methotrexate, azathioprine, tocilizumab, abatacept, leflunomide, tacrolimus, tofacitinib and cyclosporine A. Participants have to be on stable monotherapy with any of these medications for at least 6 months prior to visit 1
  19. Combined therapy of two or more of the following therapeutics: mycophenolate mofetil/sodium, methotrexate, azathioprine, tocilizumab, abatacept, leflunomide, tacrolimus, tofacitinib and ciclosporine A within at least 8 weeks prior to visit 1.
  20. Need for full-dose therapeutic anticoagulation (e.g. vitamin K antagonists, direct thrombin inhibitors or heparin)
  21. Previous hematopoietic stem cell transplantation (HSCT) within 12 months of Visit 1, or HSCT planned within 12 months after Visit 1.
  22. Other investigational therapy received within 1 month or 6 half-lives (whichever was greater) prior to screening visit.

      Prior/Concurrent Clinical Study Experience
  23. Prior participation in FMT study in the last 12 months. Diagnostic assessments
  24. Abnormal coagulation parameters as defined as International normalised ratio (INR) >2, prolongation of prothrombin time (PT) and partial thromboplastin time (PTT) by >1.5 x ULN at Visit 1 Other Exclusions
  25. Women who are pregnant, nursing, or who plan to become pregnant while in the trial. (Women of child bearing potential should be tested with Hcg (urine or serum). Woman of child bearing potential if not using highly efficient contraception.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2020-09-24 (Actual); Primary Completion 2022-06-27 (Actual); Study Completion 2022-06-27 (Actual)

PRIMARY OUTCOMES:
• Change from baseline to week 12 in UCLA GIT score item diarrhea or bloating, depending which was the worst symptom at baseline evaluated separately for each patient | baseline to week 12
  The UCLA GIT score is a validated patient reported outcome measure capturing and grading GI symptoms related to SSc. The bloating scale is scored on a Visual Analog Scale from 0 (better) to 3 (worse) and the diarrhea scale from 0 (better) to 2.5 (worse). Change=(week12 score-baseline score)

SECONDARY OUTCOMES:
• Safety and tolerability assessed by adverse event (AE) monitoring, physical examination and clinical laboratory testing from baseline to the end of the study period | • Over the study period of 20 (+16) weeks
  • Registration of number of adverse events adverse event (AE), assessment of physical examination and clinical laboratory testing by standardized assessments and sampling
• Change from baseline to week 12 in total UCLA GIT score | baseline, week 6 and week 12.
  The UCLA GIT score is a validated patient reported outcome measure capturing and grading GI symptoms related to SSc. The total scale is scored on a Visual Analog Scale from 0 (better) to 3 (worse). Change=(week12 score-baseline score)
• Change from baseline to week 12 in UCLA GIT score item diarrhea | baseline to week 12
  The UCLA GIT score is a validated patient reported outcome measure capturing and grading GI symptoms related to SSc. The diarrhea scale is scored on a Visual Analog Scale from 0 (better) to 2.5 (worse) . Change=(week12 score-baseline score)
• Change from baseline to week 12 in UCLA GIT score item bloating | baseline to week 12
  The UCLA GIT score is a validated patient reported outcome measure capturing and grading GI symptoms related to SSc. The bloating scale is scored on a Visual Analog Scale from 0 (better) to 3 (worse) . Change=(week12 score-baseline score)

OTHER OUTCOMES:
• Change from baseline to week 12 in Faecal incontinence quality of life scale | baseline to weeks 12
  Fecal Incontinence Quality-of-Life Scale is a validated patients reported outcome divided in four subscales all rated from 1-4 (5,6) by 1 having lowest quality of life. Change=(week12 score-baseline score)
• Change from baseline to week 12 in UCLA GIT score item reflux | baseline to week 12
  The UCLA GIT score is a validated patient reported outcome measure capturing and grading GI symptoms related to SSc. The reflux scale is scored on a Visual Analog Scale from 0 (better) to 3 (worse) . Change=(week12 score-baseline score)
• Change from baseline to week 12 in UCLA GIT score item fecal soilage | baseline to week 12
  The UCLA GIT score is a validated patient reported outcome measure capturing and grading GI symptoms related to SSc. The fecal soilage scale is scored on a Visual Analog Scale from 0 (better) to 3 (worse) . Change=(week12 score-baseline score)
• Change from baseline to week 12 in UCLA GIT score item constipation | baseline to week 12
  The UCLA GIT score is a validated patient reported outcome measure capturing and grading GI symptoms related to SSc. The constipation scale is scored on a Visual Analog Scale from 0 (better) to 2.5 (worse) . Change=(week12 score-baseline score)
• Change from baseline to week 12 in UCLA GIT score item emotional wellbeing | baseline to week 12
  The UCLA GIT score is a validated patient reported outcome measure capturing and grading GI symptoms related to SSc. The emotional wellbeing scale is scored on a Visual Analog Scale from 0 (better) to 3 (worse) . Change=(week12 score-baseline score)
• Change from baseline to week 12 in UCLA GIT score item social participation | baseline to week 12
  The UCLA GIT score is a validated patient reported outcome measure capturing and grading GI symptoms related to SSc. The social participation scale is scored on a Visual Analog Scale from 0 (better) to 3 (worse) . Change=(week12 score-baseline score)
• Change from baseline to week 12 in • Change from baseline to week 12 in HAQ-DI scores | baseline to week 12
  The HAQ-DI is a patient reported outcome measuring generic health status and quality of life scale ranging from 0 to 3, with no difficultie (scale 0) up to major difficulties (scale 3). Change=(week12 score-baseline score)
• Change from baseline to week 12 in VAS Fatigue scale | baseline to week 12
  The fatigue scale measures fatigue representing how the participant feel, along a visual analogue line that extends between "not at all tired" (0) to "extremely tired" (10). Change=(week12 score-baseline score)
• Change from baseline to week 12 in ScleroId score | baseline to week 12
  The ScleroId has 10 SSc specific questionnes all along a visual analogue line that extends between "none" (0) to "extreme" (10) with a maximum score of 100. Change=(week12 score-baseline score)
• Change from baseline to weeks 2, 6 and 12 in overall faecal microbiome composition measured by 16sRNA based methods | baseline to week 2, 6 and 12
  16sRNA based methods measure the fecal microbiota composition and will be assessed at 4 timepoints. Changes from baseline to week 2,6 and 12 will be assessed.
• Change from baseline to week 12 in saliva, skin and urine microbiome measured by 16sRNA based methods | baseline to week 12
  16sRNA based methods measure the microbiota composition and will be assessed at 4 timepoints. Changes from baseline to week 2,6 and 12 will be assessed.
• Change from baseline to weeks 2, 6 and 12 in immunoglobulin bound fraction of the overall faecal microbiome | • Baseline up to week 2, 6 and 12
  16sRNA based methods measure the fecal microbiota composition which is Ig coated and will be assessed at 4 timepoints. Changes from baseline to week 2,6 and 12 will be assessed.
• Change from baseline to week 12 in gastrointestinal transit time and contractions evaluated by SmartPill technology along with registration of stool frequency and consistency by Bristol Stool Scale | Baseline to week week 12
  In a subgroup of patients SmartPill technology assesses gastrointestinal transit time. Chenges will be assessed frombaseline to week 12
• Change from baseline to weeks 6 and 12 in peripheral blood B cell and T cells (as evaluated by receptor sequencing, proteomics and cellular phenotyping) and content of soluble molecules | baseline to week 6 and 12
  Blood samples will be assessed for changes from baseline to weeks 6 and 12
• Change from baseline to weeks 2 and 12 in the architecture and cellular composition of duodenal biopsy specimens (including characterization of cellular surface markers, proteomics, metabolomics and immune cell receptor sequencing | Baseline to week 2 and 12
  Tissue samples will be assessed from skin and intestines and changes from baseline to weeks 2 and 12 determined
• Change from baseline to week 12 in skin properties evaluated by elastography and ultrasonographic skin thickness | week 12 to week 12
  Elastography assess skin properties and will be assessed in a subset of patients at baseline and week 12
• Change from baseline to week 12 in Health-related Quality of Life assessed by EQ-5D | baseline to week 12
  The EQ-5D is a generic health status and quality of life scale. The respondents evaluate their overall health status using the visual analogue scalend scales of 1-3 with higher values having worse health. Change=(week12 score-baseline score)
• Change from week 12 through week 20 in all participants, and up to week 36 in a subset of participants in UCLA GIT score item diarrhea or bloating, depending which was the worst symptom at the baseline evaluated separately for each patient | week 12 to 20 and 36
  The UCLA GIT score is a validated patient reported outcome measure capturing and grading GI symptoms related to SSc. The diarrhea scale is scored on a Visual Analog Scale from 0 (better) to 2.5 (worse), the bloting from 0-3. Change=(week20 score-week 12 score)
• Follow changes of UCLA total GIT score from week 12 through week 20 in all participants, and up to week 36 in a subset of participants | week 12 to 20 and 36
  The UCLA GIT score is a validated patient reported outcome measure capturing and grading GI symptoms related to SSc. The total scale is scored on a Visual Analog Scale from 0 (better) to 3 (worse). Change=(week20 score-week 12 score)
• Follow changes in mean of HAQ-DI; VAS Fatigue; ScleroId score; and patient reported global assessment from week 12 through week 20 in all participants, and up to week 36 in a subset of participants | week 12 to 20 and 36
  See endpoints explained above for the different outcome measures and explanations
• Assess changes of overall faecal microbiome composition measured by 16sRNA based methods from week 12 through week 20 in all participants, and up to week 36 in a subset of participants | week 12 to 20 and 36
  16sRNA based methods measure the microbiota composition and will be assessed at week 12, 20 and partly 36. Changes from to week 12 to week 20 and in a subset to week 36 will be assessed.
• Assess change of saliva, skin and urine microbiome measured by 16sRNA based methods from week 12 through week 20 in all participants | week 12 to 20
  16sRNA based methods measure the microbiota composition and will be assessed at week 12 and 20. Changes from week 12 to week 20 will be assessed.
• Assess change in peripheral blood B cell and T cells and content of soluble molecules from week 12 through week 20 in all participants, and up to week 36 in a subset of participants | week 12 to 20 and 36
  Blood samples will be assessed for changes from week 12 to week 20 and 36 in a subset
• Assess changes in upper GIT scores from week 12 to 20 and determine potential associations to the architecture and cellular composition of oesophagus biopsy specimens | week 12 to 20
  The UCLA GIT score is a validated patient reported outcome measure capturing and grading GI symptoms related to SSc. The reflux scale is scored on a Visual Analog Scale from 0 (better) to 3 (worse) . Change=(week20 score-week 12 score) and assess changes in association with øsophagus biopsies
• Assess change from week 12 to 20 in Health-related Quality of Life assessed by EQ-5D from week 12 through week 20 in all participants, and up to week 36 in a subset of participants | week 12 to 20 and 36
  The EQ-5D is a generic health status and quality of life scale. The respondents evaluate their overall health status using the visual analogue scalend scales of 1-3 with higher values having worse health. Change=(week20 and 36 score-week 12 score)

CONTACTS AND LOCATIONS:
Overall Officials: Anna-Maria Hoffmann-Vold, MD, PhD, Principal Investigator — Oslo University Hospital
Locations (4):
- Norway (4):
  - Haukeland University Hospital, Bergen
  - Oslo University Hospital, Oslo
  - University hospital of North Norway, Tromsø
  - St. Olavs hospital, Trondheim university hospital, Trondheim

IPD SHARING:
Plan to Share IPD: Yes
The investigators plan to publish the protocol and statistical analysis plan separately. The IPD will be published according to relevant legislation and as required by publishing authority.
Supporting Information: Study Protocol, SAP
Time Frame: Not known yet.
Access Criteria: Not known yet.

REFERENCES:
- [Background] Kowal-Bielecka O, Fransen J, Avouac J, Becker M, Kulak A, Allanore Y, Distler O, Clements P, Cutolo M, Czirjak L, Damjanov N, Del Galdo F, Denton CP, Distler JHW, Foeldvari I, Figelstone K, Frerix M, Furst DE, Guiducci S, Hunzelmann N, Khanna D, Matucci-Cerinic M, Herrick AL, van den Hoogen F, van Laar JM, Riemekasten G, Silver R, Smith V, Sulli A, Tarner I, Tyndall A, Welling J, Wigley F, Valentini G, Walker UA, Zulian F, Muller-Ladner U; EUSTAR Coauthors. Update of EULAR recommendations for the treatment of systemic sclerosis. Ann Rheum Dis. 2017 Aug;76(8):1327-1339. doi: 10.1136/annrheumdis-2016-209909. Epub 2016 Nov 9. PMID 27941129
- [Background] Hansi N, Thoua N, Carulli M, Chakravarty K, Lal S, Smyth A, Herrick A, Ogunbiyi O, Shaffer J, Mclaughlin J, Denton C, Ong V, Emmanuel AV, Murray CD. Consensus best practice pathway of the UK scleroderma study group: gastrointestinal manifestations of systemic sclerosis. Clin Exp Rheumatol. 2014 Nov-Dec;32(6 Suppl 86):S-214-21. Epub 2014 Nov 5. PMID 25372804
- [Background] Volkmann ER, Hoffmann-Vold AM, Chang YL, Jacobs JP, Tillisch K, Mayer EA, Clements PJ, Hov JR, Kummen M, Midtvedt O, Lagishetty V, Chang L, Labus JS, Molberg O, Braun J. Systemic sclerosis is associated with specific alterations in gastrointestinal microbiota in two independent cohorts. BMJ Open Gastroenterol. 2017 Apr 1;4(1):e000134. doi: 10.1136/bmjgast-2017-000134. eCollection 2017. PMID 28761687
- [Background] van Nood E, Vrieze A, Nieuwdorp M, Fuentes S, Zoetendal EG, de Vos WM, Visser CE, Kuijper EJ, Bartelsman JF, Tijssen JG, Speelman P, Dijkgraaf MG, Keller JJ. Duodenal infusion of donor feces for recurrent Clostridium difficile. N Engl J Med. 2013 Jan 31;368(5):407-15. doi: 10.1056/NEJMoa1205037. Epub 2013 Jan 16. PMID 23323867
- [Background] Staley C, Kaiser T, Vaughn BP, Graiziger C, Hamilton MJ, Kabage AJ, Khoruts A, Sadowsky MJ. Durable Long-Term Bacterial Engraftment following Encapsulated Fecal Microbiota Transplantation To Treat Clostridium difficile Infection. mBio. 2019 Jul 23;10(4):e01586-19. doi: 10.1128/mBio.01586-19. PMID 31337728
- [Background] Juul FE, Garborg K, Bretthauer M, Skudal H, Oines MN, Wiig H, Rose O, Seip B, Lamont JT, Midtvedt T, Valeur J, Kalager M, Holme O, Helsingen L, Loberg M, Adami HO. Fecal Microbiota Transplantation for Primary Clostridium difficile Infection. N Engl J Med. 2018 Jun 28;378(26):2535-2536. doi: 10.1056/NEJMc1803103. Epub 2018 Jun 2. No abstract available. PMID 29860912
- [Background] Khanna D, Hays RD, Maranian P, Seibold JR, Impens A, Mayes MD, Clements PJ, Getzug T, Fathi N, Bechtel A, Furst DE. Reliability and validity of the University of California, Los Angeles Scleroderma Clinical Trial Consortium Gastrointestinal Tract Instrument. Arthritis Rheum. 2009 Sep 15;61(9):1257-63. doi: 10.1002/art.24730. PMID 19714600
- [Background] Khanna D, Furst DE, Maranian P, Seibold JR, Impens A, Mayes MD, Clements PJ, Getzug T, Hays RD. Minimally important differences of the UCLA Scleroderma Clinical Trial Consortium Gastrointestinal Tract Instrument. J Rheumatol. 2011 Sep;38(9):1920-4. doi: 10.3899/jrheum.110225. Epub 2011 Jul 1. PMID 21724699
- [Background] Dehli T, Martinussen M, Mevik K, Stordahl A, Sahlin Y, Lindsetmo RO, Vonen B. Translation and validation of the Norwegian version of the fecal incontinence quality-of-life scale. Scand J Surg. 2011;100(3):190-5. doi: 10.1177/145749691110000310. PMID 22108748
- [Background] Yang Y, Qiu L, Wang L, Xiang X, Tang Y, Li H, Yan F. Quantitative Assessment of Skin Stiffness Using Ultrasound Shear Wave Elastography in Systemic Sclerosis. Ultrasound Med Biol. 2019 Apr;45(4):902-912. doi: 10.1016/j.ultrasmedbio.2018.11.015. Epub 2019 Jan 18. PMID 30665723
- [Background] Benno P, Norin E, Midtvedt T, Hellstrom PM. Therapeutic potential of an anaerobic cultured human intestinal microbiota, ACHIM, for treatment of IBS. Best Pract Res Clin Gastroenterol. 2019 Jun-Aug;40-41:101607. doi: 10.1016/j.bpg.2019.03.003. Epub 2019 Apr 29. PMID 31594647
- [Background] Jorup-Ronstrom C, Hakanson A, Sandell S, Edvinsson O, Midtvedt T, Persson AK, Norin E. Fecal transplant against relapsing Clostridium difficile-associated diarrhea in 32 patients. Scand J Gastroenterol. 2012 May;47(5):548-52. doi: 10.3109/00365521.2012.672587. Epub 2012 Apr 2. PMID 22468996
- [Derived] Fretheim H, Barua I, Bakland G, Dhainaut A, Halse AK, Carstens MN, Didriksen H, Midtvedt O, Lundin KEA, Aabakken L, Sarna VK, Zare HK, Khanna D, Distler O, Midtvedt T, Baekkevold ES, Olsen IC, Domanska D, Pesonen ME, Molberg O, Hoffmann-Vold AM. Faecal microbiota transplantation in patients with systemic sclerosis and lower gastrointestinal tract symptoms in Norway (ReSScue): a phase 2, randomised, double-blind, placebo-controlled trial. Lancet Rheumatol. 2025 May;7(5):e323-e332. doi: 10.1016/S2665-9913(24)00334-5. Epub 2025 Jan 31. PMID 39900089
- [Derived] Hoffmann-Vold AM, Fretheim HH, Sarna VK, Barua I, Carstens MN, Distler O, Khanna D, Volkmann ER, Midtvedt O, Didriksen H, Dhainaut A, Halse AK, Bakland G, Pesonen M, Olsen I, Molberg O. Safety and efficacy of faecal microbiota transplantation by Anaerobic Cultivated Human Intestinal Microbiome (ACHIM) in patients with systemic sclerosis: study protocol for the randomised controlled phase II ReSScue trial. BMJ Open. 2021 Jun 24;11(6):e048541. doi: 10.1136/bmjopen-2020-048541. PMID 34168032